CLINICAL TRIAL: NCT02166060
Title: Ivabradine in Patients With an Unsatisfactory Percentage of Cardiac Resynchronization Therapy
Acronym: IvaCRT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Marcin Grabowski, PhD, Medical University of Warsaw
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IvaCRT KB/111/2014
Record Dates: First submitted 2014-06-10; First posted 2014-06-18 (Estimated); Last update posted 2014-06-18 (Estimated); Status verified 2014-06

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Ivabradine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ivabradine (Experimental): Ivabradine 5 mg twice a day or 7,5 mg twice a day
  Interventions: Drug: Ivabradine

INTERVENTIONS:
Drug: Ivabradine — Ivabradine 5 mg twice a day or 7,5 mg twice a day
  Other Names: Procoralan

SUMMARY:
The purpose of this study is to determine the role of ivabradine in cardiac resynchronization recipients with an unsatisfactory percentage biventricular pacing.

The study protocol 60 patients with heart failure NYHA (New York Heart Association) II-IV treated with optimal medical therapy as clinically indicated who received CRT-D device more than 3 months ago. Patients with biventricular pacing <95% will and heart rate <70 at rest and >50% of heart rate in device memory >70 will receive ivabradine. The minimal follow-up of patients in the study will be at least six months.

DETAILED DESCRIPTION:
Approximately 30% of CRT recipients do not respond to therapy. One of the causes ot that is unsatisfactory percentage of biventricular pacing. Patients may loose biventricular pacing because of inadequate sinus tachycardia.

Ivabradine may prevent inadequate sinus tachycardia and improve quality of live of CRT recipients.

According to current guidelines ivabradine is recommended in patients with symptomatic heart failure with heart rate at rest >70.

The hypothesis of this study is that ivabradine may increase percentage of biventricular pacing in CRT recipients who have unsatisfactory percentage of biventricular pacing and >50% of heart rate in device memory >70.

ELIGIBILITY:
Inclusion Criteria:

* heart failure NYHA II-IV
* left ventricular ejection fraction =<35%
* CRT-D implanted over 3 months ago
* optimal CRT-D parameters
* biventricular pacing <95% despite the optimal parameters of the device
* optimal pharmacotherapy with the highest well-tolerated beta-adrenolytic dosage
* heart rate at rest below 70 bpm
* over 50% of heart rhythm over 70 bpm at interrogation with the device

Exclusion Criteria:

* persistent atrial fibrillation/flutter
* device associated ineffective resynchronization
* contraindications to ivabradine

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-08; Primary Completion 2016-08 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Percentage of biventricular pacing >95% | 6 months

SECONDARY OUTCOMES:
Percentage of biventricular pacing >98% | 6 months
Time to first inappropriate shock | 6 months
change of mean heart rate compared with baseline | 6 months
Cardiovascular hospitalization | 6 months
The change between baseline and final echocardiographic parameters | 6 months
The assessment of quality of life (SF36) | 6 months
The change between baseline and final NYHA class | 6 months

OTHER OUTCOMES:
Number of participants with adverse events | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Marcin Grabowski, MD, Study Chair — Medical University of Warsaw
Locations (1):
- 1st Department of Cariology of Medcial University of Warsaw, Warsaw, Masovian Voivodeship, Poland